CLINICAL TRIAL: NCT02459249
Title: Treatment of Metabolic Alterations in Adults Living in Communities With Low Socioeconomic Status
Brief Title: Metabolic Syndrome Diagnosis and Treatment for Adults of Low Socioeconomic Status Communities
Acronym: PrEVEnTYCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Ismael Campos, Doctor, researcher, Mexican National Institute of Public Health
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1206-6941 CI:1198
Record Dates: First submitted 2015-04-06; First posted 2015-06-02 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; High Blood Pressure; Hyperglycemia; Dyslipidemia
MeSH Terms: conditions — Obesity; Hypertension; Hyperglycemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Lifestyle (Experimental): A physician and a nutritionist will be give recommendations for diet and exercise emphasizing the importance of a healthy lifestyle (suggesting moderate-intensity activity at least 150 minutes/week and to eat less sodium, fat, sugar, portions and calories). Verbal and written individualized recommendations from trained professionals (nutritionists, and physician) will be provided. Monthly sessions of at least 30 minutes covering diet, exercise, and behavior modifications were held. The first was a one-to-one meeting and was followed by group sessions based on behavioral counseling
  Interventions: Other: Healthy Lifestyle
- Treatment of Mexican Health Minister (Placebo Comparator): General and unspecific recommendations of diet and physical activity for the metabolic syndrome treatment, given for a physician
  Interventions: Other: Placebo Comparator (Treatment of Mexican Health Minister)

INTERVENTIONS:
Other: Healthy Lifestyle — A physician and a nutritionist will be give recommendations for diet and exercise emphasizing the importance of a healthy lifestyle (suggesting moderate-intensity activity at least 150 minutes/week and to eat less sodium, fat, sugar, portions and calories). Verbal and written individualized recommendations from trained professionals (nutritionists, and physician) will be provided. Monthly sessions of at least 30 minutes covering diet, exercise, and behavior modifications were held. The first was a one-to-one meeting and was followed by group sessions based on behavioral counseling
  Arms: Healthy Lifestyle
Other: Placebo Comparator (Treatment of Mexican Health Minister) — General and unspecific recommendations of diet and physical activity for the metabolic syndrome treatment, given for a physician
  Arms: Treatment of Mexican Health Minister

SUMMARY:
The objective of this study is to evaluate the effect of a healthy-habits intervention tailored to the cultural, economical and social context of the target population in cardiometabolic parameters, for a population with no access to specialized health services. The intervention was designed considering environmental and economic context like availability of food and physical activity spaces; cultural factors like social and culinary traditions; individual food preferences. It encompass a selected set of behavioral and nutritional strategies aiming to achieve control of metabolic disorders involved and to reduce the risk for diabetes.

The investigators' study is a nine-month clinical intervention with randomized allocation, and parallel assignment. For the first six months, the participants in the control group will receive the treatment from the primary care service by the Health Minister as implemented by the local health center, and for the intervention group participants will receive a treatment to improve the quality of the diet and promote the practice of physical activity. Both groups will be reevaluated at third, sixth and ninth-months follow-up. The physician and the nutritionist of the study will be give the recommendations for diet and advice on exercise, mainly by suggesting moderate-intensity activity, such as brisk walks for at least 150 minutes/week.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of a low-cost healthy-habits intervention tailored to the cultural, economical and social context of the target population in cardiometabolic parameters , for a population with no access to specialized health services. The intervention was designed considering environmental and economic context like availability of food and physical activity spaces; cultural factors like social and culinary traditions; individual food preferences. It encompass a selected set of behavioral and nutritional strategies aiming to achieve control of metabolic disorders involved and to reduce the risk for diabetes.

MATERIAL AND METHODS:

The investigators' study is a nine-month clinical intervention with randomized allocation, and parallel assignment. For the first six months, the participants in the control group will receive the treatment from the primary care service by the Health Minister (Treatment protocols for the components of the metabolic syndrome) as implemented by the local health center, and for the intervention group participants will receive a treatment to improve the quality of the diet and promote the practice of physical activity. Both groups will be reevaluated at third, sixth and ninth-months follow-up. The physician and the nutritionist of the study will be give the recommendations for diet and advice on exercise, mainly by suggesting moderate-intensity activity, such as brisk walks for at least 150 minutes/week.

For the diagnosis of MS, the investigators used the classification from the International Diabetes Federation, and therefore participants were required to have three or more of the following criteria: a) waist circumference ≥ 90 cm in men and ≥ 80 cm in women, b) triglycerides ≥150 mg/dL, c) high density lipoprotein (HDL-cholesterol) < 40 mg/dL in men and < 50 mg/dL in women, d) blood pressure ≥130/85 mmHg; and e) fasting glucose ≥100 mg/dL.

Sample Size. Power size was estimated assuming a 2-sided t-test with an alpha of 0.05 and a power of 80%. Data for the estimation (standard deviation, expected mean difference in indicators) were taken from a previous study on similar population. The investigators expect a difference in prevalence of MS components of at least 10 prevalence points, (-5% control, -10% intervention groups). The sample size was 60 persons per experimental condition (total = 120).

Recruitment:

The study was conducted in a rural county of central Mexico. Individuals were invited to participate in a screening for MS through postings in public areas and using traditional social networks. During screening, individuals interested in participating received an explanation of the study. Upon agreement trained and standardized personnel took their medical history, anthropometric measurements (weight, height, and waist circumference) blood pressure and venous blood samples for determination of glucose, triglycerides, and HDL-cholesterol. The first 120 candidates will be accepted to the study. In addition to the criteria already mentioned, the investigators will record the address of the candidates, so the investigators can identify if two or more live in the same household.

Randomization Participants will be randomly allocated by matched pairs. The variables of matching are: in-house social support (whether or not there is another person interested in changing lifestyles in the household), and level of self-efficacy to follow the structured diet. Then, within matched pairs, the investigators will randomly allocate the treatment condition.

Study Procedures:

The intervention group received general information from a physician of the study, emphasizing the importance of a healthy lifestyle. Verbal and written individualized recommendations from trained professionals (nutritionists, and physician) will be provided. From first month to six month, monthly sessions of at least 30 minutes covering diet, exercise, and behavior modifications were held. The first was a one-to-one meeting and was followed by group sessions based on behavioral counseling (Explanations about benefits of diet and exercise in controlling metabolic abnormalities) and healthy habits tips

During the sessions, an individually prescribed diet was given, in line with existing guidelines. Similarly, advice on exercise was given, mainly by suggesting moderate-intensity activity, such as brisk walks for at least 150 minutes/week.

The control group with treatment from the primary care service received specific individualized programs.

Both groups will be reevaluate at zero, three and six months follow-up.

Intervention Development:

The intervention is psychologically based on the transtheoretical model of change and the theory of self-regulation. A review of evidence-based practices for short and long-term weight loss was also performed, yielding similar conclusions as those from professional review panels. The psychological processes that the investigators aim to influence with the intervention were: social support, feedback and self-monitoring, counterconditioning, goal setting, and stimuli control. For each process, the investigators developed an intervention component. The development of these components was based on an iterative methodology and a human-centered approach, which is described in more detail in another paper. The development of the intervention components was done using a design thinking approach. Through an iterative process that mixed the development of prototypes with collection of data regarding the context and the target population, the researchers progressively refined the investigators' intervention components.

Structured diet. Starting with a physiologically based model, the investigators developed multiple prototypes, aiming to satisfy not only nutritional requirements but also population constrains, such as food cost, availability and skills. Finally, the investigators adapted the menus to the culinary traditions of the target population.

Skills Workshops. Formative research yielded that the most important food behaviors that were necessary to work on were processed food skills, cooking skills and social support skills.

Goal setting. A commitment contract will be provided to. participants. They will be invited to define monthly goals in terms of health parameters or appearance (to be fit or slim), in accordance with their clinical plans These contracts are with themselves or significant others and can have small rewards. The only requirement is that the goals are approved by clinicians and the contracts promote adherence to treatment.

Feedback component. A food journaling tool will be provided to participants. They will be invited to follow a food and physical activity journal, along with weight measurement daily or every other day. For participants with low literacy levels, the investigators will provide a plate or container to help with measurement. In addition, the results of physiological test will be provided right away, so they know how far they are of their goals.

Stimuli Control. A workshop regarding on how to reshape their food environments at home and at work will be given, so the adherence to the lifestyles changes becomes easier.

Household social-support: a workshop aimed to improve participants ability to negotiate social support will be provided. They were encouraged to obtain a "partner in lifestyle or physical appearance challenge" in their household. This partner was able to assist more in the same workshops and consultations than the main participant.

Analysis. To evaluate the effect of the intervention, the investigators will utilize a structural causal model (SCM). The target causal parameter of interest is the effect of the intervention in the prevalence of MS components, the average treatment effect of the experimental intervention. The investigators commit to use an estimate based on the G-comp formula. The investigators will assess positivity assumptions prior to analysis and adjust for practical violations of it. The investigators will test different estimation methods for this target estimate (ATE), including both parametric and non-parametric. The investigators will use a preestablished set of methods and a criteria to choose among them (most likely the lossless function). This method, called super learner, is described in further detail in (Van der Laan, Petersen).

The investigators will estimate both the average treatment effect (ATE) and the conditional treatment effect (cTE).

Ethical approval. The study was conducted with approval of the Ethics and Research Committees at the National Institute of Public Health, Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 20-55 years old with MS,
* without access to specialized health services,
* residents in rural communities of the state of Morelos-Mexico,
* and without current treatment for MS

Exclusion Criteria:

* Having bariatric surgery for weight loss,
* current treatment for MS,
* hypothyroidism,
* cancer,
* smoking,
* use of alcohol or drugs,
* psychiatric disorders,
* anti-obesity medication,
* women using birth control methods, pregnant, lactating or near menopause,
* body weight gain or loss greater than two percent two months prior to the start of the study and
* pharmacological treatment for diabetes (or fasting glucose ≥300 mg/dL); hypertension (or ≥150/110 mmHg); or dyslipidaemia (triglycerides ≥400 mg/dL).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Metabolic Syndrome | Baseline
Number of Participants with Metabolic Syndrome | 3 months
Number of Participants with Metabolic Syndrome | 6 months
Number of Participants with Metabolic Syndrome | 9 months

SECONDARY OUTCOMES:
Changes in body weight | 3 months
Changes in body weight | 6 months
Changes in body weight | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ismael R Campos, PhD, Study Director — National Institute of public Health
Locations (1):
- National Institute of Public Health, Cuernavaca, Morelos, Mexico